CLINICAL TRIAL: NCT00701493
Title: An Open-Label, Randomized, 2-Way Crossover Study of the Bioavailability of an Oral Liquid Formulation Relative to the Marketed Sprinkle Capsule Formulation of Topiramate RWJ-17021-000 in Healthy Subjects
Brief Title: A Phase 1 Bioavailability Study of Topiramate Oral Liquid Formulation Compared to the Marketed Sprinkle Capsule Formulation in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR002239
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Epilepsy
Keywords: Topiramate; Topiramate oral liquid; TOPAMAX Sprinkle capsule; topiramate capsules
MeSH Terms: conditions — Epilepsy

INTERVENTIONS:
Drug: Topiramate oral liquid formulation;Topiramate Sprinkle formulation

SUMMARY:
The primary purpose of this study is to estimate the bioavailability of the oral liquid formulation of topiramate relative to the commercially available oral sprinkle capsule formulation in healthy patients. If appropriate, bioequivalence between the oral liquid formulation and the sprinkle capsule formulation will be assessed.

DETAILED DESCRIPTION:
This is a randomized, open-label, 2-way crossover, single-center, relative bioavailability study in healthy adult men and women. The study was conducted in 3 phases: a pretreatment phase (Days -14 to -1), a 25-day open-label treatment phase, and a 7-day follow-up phase. Patients will enter the screening phase no more than 14 days prior to receiving study treatment. During the screening period, patients' eligibility will be assessed, and physical examinations and other safety evaluations will be performed. Eligible patients will be randomized at baseline (Day -1) to receive the topiramate oral liquid and sprinkle capsule formulations according to 1 of 2 treatment sequences (see Section 5, Randomization and Blinding). There will be a 3 week washout period between treatments. Initially, approximately 40 patients will be enrolled in the study, in order for at least 32 patients to complete all PK assessments. Patient will be confined to the study site on the evenings of Days -1 and 20. Following a 10-hour overnight fast, patients will receive topiramate as a single 100-mg dose of the oral liquid formulation and the oral sprinkle capsule formulation according to the sequence specified by the randomization schedule at approximately 8 a.m. on Days 1 and 21. Serial blood samples will be collected for estimation of plasma topiramate concentrations at scheduled times from predose through 96 hours postdose. Patients will be discharged from the study site on Days 3 and 23 after collection of the 48 hour postdose blood sample. Patients will arrive at the study site 2 hours prior to PK sample collection to obtain the 60 hour (Days 3 and 23), 76 hour (Days 4 and 24), and 96 hour (Days 5 and 25) postdose samples. Patients will complete the study on Day 25 and receive a follow-up phone call on Day 32 for an adverse event assessment. Safety and tolerability will be assessed throughout the study. Patients will be randomly assigned to receive both oral treatments: A then B, or B then A. Treatment A: Topiramate 100 mg as 20 mL of a 5 mg/mL liquid formulation and Treatment B: Topiramate 100 mg as 4 X 25-mg sprinkle capsule formulation There is a 3 week wash-out period between treatments

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 19 and 32 kg/m2, inclusive
* Women of non-child-bearing potential or practicing birth control
* Have a normal electrocardiogram (ECG)
* Be in good health, in the opinion of the investigator
* Be sufficiently alert to understand and communicate intelligibly with the study staff (i.e., patients must be able to perform all study procedures)
* Agree to limit their methylxanthine consumption throughout the study to 2 methylxanthine-containing substances
* Agree to refrain from ingesting products containing grapefruit, quinine, or Seville orange during the study
* Agree to refrain from ingesting antacids during the study
* Agree to refrain from ingesting alcohol during the study
* Have signed an informed consent document indicating that the study has been explained to them and they are willing to participate in the study.

Exclusion Criteria:

* History of significant renal, hepatic, gastrointestinal, hematologic, pulmonary, metabolic, thyroid, or other chronic disease
* Significant cardiovascular disease, including a history of myocardial infarction within the past 2 years, cerebrovascular accident, clinically significant cardiac valvular disease, unstable angina, significantly abnormal ECG, arrhythmia, or congestive cardiac failure
* History of significant psychiatric disorders including schizophrenia, psychosis, panic disorder, major depression, suicidal attempt or other major affective disorders or current dysthymia. If possible, the investigator shall attempt to confirm the presence or absence of past psychiatric history with subject's primary care physician
* History of raised intraocular pressure, glaucoma, or otherwise at risk for acute narrow-angle glaucoma
* Demonstrate significant active physical disease, acute or chronic, within 7 days before the start of the study
* Liver enzymes (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) outside the normal limits
* Women who wish to become pregnant within 2 months following discontinuation of the study drug, or who are breast-feeding
* Require or have taken any prescription medications within 2 weeks before dosing
* Use of any over-the-counter medications (including aspirin, antacids, vitamins, and herbal supplements (e.g., diuretic tea that may have an impact on renal function) within 7 days before dosing until the end of the study
* Use of hormonal contraceptives (including oral, implanted, intrauterine device, and patch) or hormonal replacement therapy within 3 months before start of screening until 2 months after study completion
* Use of a carbonic anhydrase inhibitor for any reason within 2 weeks before the start of screening
* History of alcohol or drug abuse
* Testing positive for HIV antibody, Hepatitis B antigen, or Hepatitis C antibody
* Abnormal clinical laboratory values, unless reviewed and approved by the Sponsor's medical monitor
* Use of any nicotine-containing products, including tobacco products (e.g., cigarettes, cigars, or chewing tobacco) in the 3 months before start of screening until the end of the study
* History of kidney stones
* Family history (first-degree relatives) of kidney stones that are not established to be due to a known cause (e.g., hyperparathyroidism, medication)
* History of lactic acidosis or chronic metabolic acidosis
* History of hereditary or acquired neurologic disease (e.g., epilepsy or significant brain trauma)
* Malignancy or a history of a malignancy within 5 years before start of screening, other than treated basal cell carcinomas of the skin
* Known contraindication or hypersensitivity to topiramate or heparin
* Use of any medications that are known P-450 enzyme inducers or inhibitors (e.g., cimetidine or rifampin), within 3 months before dosing. (See Attachment 6, Listing of Medications That Are Known Cytochrome P-450 Enzyme Inducers or Inhibitors)
* Any significant condition that in the opinion of the investigator could interfere in the patient's participation or completion of the study
* Have received an experimental drug or used an experimental medical device within 30 days before screening
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
AUClast, AUC¥, and Cmax (Area Under the Curve (last), Area Under the Curve (infinity) and maximum plasma concentration); Incidence, severity, and type of adverse event changes in laboratory results, physical exam, ECG, vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open-Label, Randomized, 2-Way Crossover Study of the Bioavailability of an Oral Liquid Formulation Relative to the Marketed Sprinkle Capsule Formulation of Topiramate RWJ-17021-000 in Healthy Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=462&filename=CR002239_CSR.pdf